CLINICAL TRIAL: NCT01453582
Title: Phase III Study of Total Flavonoids of Propolis Dropping Pill in Angina Pectoris: A Randomized, Double-Blind, Placebo-Controlled Multi-Centered Clinical Trial on Efficacy and Safety.
Brief Title: Efficacy and Safety Study of Total Flavonoids of Propolis Dropping Pill to Treat Angina Pectoris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Greenvalley Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FJ2011-1.1
Record Dates: First submitted 2011-10-13; First posted 2011-10-18 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2017-12

CONDITIONS: Stable Angina Pectoris
Keywords: Chest stuffiness of TCM; Qi deficiency and blood stasis of TCM
MeSH Terms: conditions — Angina, Stable

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propolis (Experimental): Total Flavonoids of Propolis dropping pill
  Interventions: Drug: Total Flavonoids of Propolis dropping pill
- Placebo (Placebo Comparator): Simulant of total Flavonoids of Propolis dropping pill
  Interventions: Drug: total Flavonoids of Propolis dropping pill

INTERVENTIONS:
Drug: Total Flavonoids of Propolis dropping pill — One pack contains 30 pills, weight 33g. One pack each time, three times a day, 14 days a course.
  Arms: Propolis
Drug: total Flavonoids of Propolis dropping pill — One pack contains 30 pills, weight 33g. One pack each time, three times a day, 14 days a course.
  Arms: Placebo

SUMMARY:
The purpose of this study is to confirm the efficacy and safety of total flavonoids of propolis dropping pill to treat angina pectoris, evaluated by total exercise time of treadmill exercise test.

ELIGIBILITY:
Inclusion Criteria:

* Class I, Class II and Class III stable angina pectoris, angina attack more than 3 times one week;
* Qi deficiency and blood stasis syndrome of Traditional Chinese Medicine;
* In resting electrocardiogram, ST-segment deviation≥0.05mv and/or T-wave inversion≥0.2mv in the leads R-wave is predominant during non-attack period, or ST-segment deviation≥0.1mv and/or T-wave inversion≥0.2mv in the leads R-wave is predominant during angina attack;
* Total exercise time of treadmill exercise test≥3 minutes.The discontinuance standard should be reached. And the difference of total exercise time between before and after run in period should ≤15%;
* Other confirmed diagnostic evidence of coronary heart disease, such as definite history of old myocardial infarction, or incomplete revascularization one year after coronary intervention therapy(residual luminal stenosis≥50%), or coronary angiography evidence(at least single vessel disease and luminal stenosis≥50%), or nuclein examination evidence, or computer tomography angiography evidence;
* Signed the informed consent form.

Exclusion Criteria:

* Chest pain caused by acute myocardial infarction(AMI), Class IV/serious angina pectoris, psychosis, serious neurosis, climacteric syndrome, hyperthyroidism, Cervical Spondylosis, gallbladder- heart syndrome, gastroesophageal reflux, hiatus hernia, aortic dissection, aortic valve disease;
* Not well controlled hypertension(systolic pressure≥160mmHg，diastolic pressure≥100mmHg), serious cardiopulmonary insufficiency, serious arrhythmia(rapid atrial fibrillation, atrial flutter, paroxysmal ventricular tachycardia, etc);
* Serious diseases of heart, lung, liver, kidney and blood;
* Allergic constitution or allergic to the components of total Flavonoids of Propolis dropping pill;
* Women during pregnancy or lactation;
* Received any major operation within 4 weeks;
* Have been in other clinical trials within 30 days;
* Using but can not withdraw anti-angina medicine as long acting nitrates;
* Not well controlled hyperglycemia;
* Not fit for this trial judged by investigator.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2011-12; Primary Completion 2014-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Improvement of total exercise time of treadmill exercise test | -2 week, 0 weeks, 12 weeks

SECONDARY OUTCOMES:
The marked effective rate of angina pectoris | -2 weeks, 0 week, 6 weeks, 12 weeks
  * Class I: No symptom or almost no symptom, decrease of angina pectoris total score ≥ 1/3；
  * Class II: No symptom or almost no symptom, decrease of angina pectoris total score ≥ 2/3；
  * Class III: Almost no symptom, decrease of angina pectoris total score ≥ 2/3, or the score decrease to the degree of Slight or Class I.
Attack times of angina pectoris | -2 weeks, 0 week, 6 weeks, 12 weeks
Pain degree of angina pectoris | -2 weeks, 0 week, 12 weeks
Duration of angina pectoris attack | -2 weeks, 0 week, 6 weeks, 12 weeks
Dose change of nitroglycerin | -2 weeks, 0 week, 6 weeks, 12 weeks
  * Withdraw: completely withdrawal after the treatment;
  * Decrease: decrement ≥50% after the treatment;
  * No change: decrement <50% after the treatment.
The main symptoms of Chinese Traditional Medicine | -2 weeks, 0 week, 6 weeks, 12 weeks
  Effect index = (total score before treatment - total score after treatment)/total score before treatment×100%
  * Cured: effect index ≥90%;
  * Marked effective: 90%> effect index ≥70%;
  * Effective: 70%> effect index ≥30%;
  * Ineffective: effect index <30%.
Score change of the Seattle Angina Questionnaire (SAQ) | 0 week, 12 weeks
Improvement of ECG | -2 weeks, 0 week, 12 weeks
  * Cured: normal or almost normal;
  * Marked effective: ST-segment deviation upturn≥0.05mV, but still abnormal, improvement of T-wave inversion of main leads ≥25%, or flate T-wave change to vertical, improved atrioventricular block or intraventricular block;
  * Effective: almost no charge;
  * Ineffective: anabatic ST-segment deviation, deeper T-wave, or flate T-wave change to inverted.
Improvement of other indexes of treadmill exercise test | -2 weeks, 0 week, 12 weeks
  metabolic equivalent, blood pressure, oxygen consumption, speed, grade.
Time to ST-segment deviation>1mm and positive symptoms appear | -2 weeks, 0 week, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lanjun Sun, Principal Investigator — Sencond Affiliated Hospital of Tianjin University of Traditional Chinese Medicine
Locations (13):
- China (13):
  - Guangdong Second Provincial Traditional Chinese Medicine Hospital, Guangzhou, Guangdong
  - Ruikang Hospital of Guangxi Traditional Chinese Medical University, Nanning, Guangxi
  - Hubei Hospital of Traditional Chinese Medicine, Wuhan, Hubei
  - The Affiliated Hospital to Changchun University of Chinese Medicine, Changchun, Jilin
  - Sencond Affiliated Hospital of Liaoning University of Traditional Chinese Medicine, Shenyang, Liaoning
  - Affiliated Hospital of Liaoning University of Traditional Chinese Medicine, Shenyang, Liaoning
  - Neimenggu Hospital of Traditional Chinese and Mongolian Medicine, Hohhot, Neimenggu
  - Shanghai Hospital of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Shuguang Hospital, Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Shanxi Hospital of Traditional Chinese Medicine, Taiyuan, Shanxi
  - Second Affiliated Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality
  - Xinjiang Hospital of Traditional Chinese Medicine, Ürümqi, Xinjiang